CLINICAL TRIAL: NCT02538016
Title: Use of Tolvaptan, a Vasopressin Antagonist, to Increase Urine Dilution and Reduce Cystine Urolithiasis Among Patients With Homozygous Cystinuria: a Pilot Investigation
Brief Title: TCUPS- Tolvaptan Use in Cystinuria and Urolithiasis: A Pilot Study
Acronym: TCUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caleb Nelson (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Caleb Nelson, MD, MPH, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16726
Record Dates: First submitted 2015-07-21; First posted 2015-09-02 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-05

CONDITIONS: Cystinuria
Keywords: Cystinuria; Kidney Stones
MeSH Terms: conditions — Cystinuria; Kidney Calculi | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolvaptan (Other)
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
The goal of this research project is to establish that in short-term use, tolvaptan is a safe and potentially effective new therapy for cystinuria, by conducting a short-term pilot study of the safety and tolerability of this drug, and assess impact on urinary stone risk parameters, among adolescent and young adult patients with clinical cystinuria.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 12 - 29 years
* Weight ≥ 25kg (55 lbs)
* Confirmed cystinuria diagnosis
* Specific blood test levels (done within the past 6 months)

Exclusion Criteria:

* Concurrent non-renal disease that might increase risk of complications due to aquaresis
* Liver or biliary disease (chronic or acute)
* Malabsorption syndrome or other gastrointestinal condition that may interfere with response to therapy
* Non-cutaneous malignancy within last 5 years
* History of adverse reaction or allergy to Tolvaptan or other arginine vasopressin V2-receptor antagonists

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caleb Nelson, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and Enrollment period was between August 2016 to December 2018. Subjects were recruited from our existing database of cystinuria patients, from new patients presenting during the research period, and via advertising through the International Cystinuria Foundation, Rare Kidney Stone Consortium, and social media.
Pre-assignment Details: Of 6 eligible and interested participants, 5 met inclusion criteria and were consented, and of these, 1 withdrew prior to travel to our hospital for drug administration.
Groups:
- Tolvaptan: This was a single arm, unblinded study. All participants received half of the recommended dose (weight-dependent) on Days 1 through 4 and then the full recommended dose (weight-dependent) on Days 5 through 8
  Example of Dosing Schedule by Weight:
  Participant Weight is between: 12.5 kg -37.49 kg Then their Dose on Days 1-4 = 7.5mg (.6mg/kg -.2mg/kg) Dose on Days 5-8 is doubled = 15mg (1.2mg/kg - .4mg/kg)
  Maximum dose administered was 60 mg.
Period: Overall Study
Arm/Group | Tolvaptan
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tolvaptan
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Urinary Cystine Supersaturation (mg/L) at High Dose (Day7-8)
Description: The primary outcome was urinary cystine supersaturation as measured by "cystine capacity". This proprietary test (Litholink Corp., Chicago IL) is reported as a value in mg/L above or below zero, with positive values indicating urine undersaturated with cystine, while negative values indicate that the urine is supersaturated with cystine. Four 24-hour urine samples were obtained during the study: one at baseline 3-6 days prior to the measurement, one on day 3-4 of the dosing period, one on day 7-8 of the dosing period, and one 3-6 days after the washout period. Each 24 hour urine sample was sent individually for analysis by Litholink Corp, which performs the cystine assays.
Time Frame: 23 days
Measure: Mean (Full Range); unit: mg/L
Groups:
- Tolvaptan: Tolvaptan.
Arm/Group | Tolvaptan
Number analyzed (Participants) | 4
mg/L | 70 [-3 to 111]

2. Secondary Outcome: Urine Osmolality at High Dose (Day 8)
Description: Secondary outcomes included serum sodium and other electrolyte levels. Serum electrolytes for each subject before, during, and after tolvaptan treatment (Sodium/Potassium/Chloride in mmol/L).
Time Frame: 11 days
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Tolvaptan
Number analyzed (Participants) | 4
mmol/L
  Sodium | 141 [139 to 142]
  Potassium | 4.05 [3.7 to 4.4]
  Chloride | 102 [101 to 103]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=4)
Severe Thirst (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02538016/Prot_SAP_000.pdf